CLINICAL TRIAL: NCT02061709
Title: A Double-Blind, Randomised, Placebo-Controlled Study to Evaluate Three Dose Regimens of Ragweed-SPIRE in Ragweed Allergic Subjects Following Challenge With Ragweed Allergen in an Environmental Exposure Chamber
Brief Title: Evaluating the Efficacy of Ragweed-SPIRE Following Exposure to Ragweed Allergen in an Environmental Exposure Chamber
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR006
Record Dates: First submitted 2014-02-03; First posted 2014-02-13 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Rhinoconjunctivitis; Rhinitis; Seasonal; Ragweed; Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ragweed-SPIRE 1 (Experimental): Ragweed SPIRE regimen 1 given 2 weeks apart
  Interventions: Biological: Ragweed-SPIRE
- Ragweed-SPIRE 2 (Experimental): Ragweed-SPIRE regimen 2 given 2 weeks apart
  Interventions: Biological: Ragweed-SPIRE
- Ragweed-SPIRE 3 (Experimental): Ragweed-SPIRE regimen 3 given 2 weeks apart
  Interventions: Biological: Ragweed-SPIRE
- Placebo (Placebo Comparator): Placebo given 2 weeks apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ragweed-SPIRE
  Arms: Ragweed-SPIRE 1; Ragweed-SPIRE 2; Ragweed-SPIRE 3
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Ragweed-SPIRE is safe and effective at reducing allergy symptoms in people who suffer from allergy to Ragweed pollen

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years.
* Reliable history consistent with moderate to severe rhinoconjunctivitis on exposure to ragweed for at least the previous two seasons.
* Minimum qualifying rhinoconjunctivitis symptom scores
* Ragweed-specific Immunoglobulin E (IgE) > 0.70 kU/L.

Exclusion Criteria:

* Subjects with a history of ragweed pollen induced asthma
* A history of anaphylaxis to ragweed allergen.
* FEV1 < 80 % of predicted.
* Subjects who cannot tolerate Baseline Challenge in the EEC.
* Subjects for whom administration of epinephrine is contraindicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).
* History of immunopathological diseases (e.g. multiple sclerosis) that in the opinion of the Investigator or the Sponsor could interfere with the results obtained from the study.
* A history of severe drug allergy, severe angioedema or anaphylactic reaction to food.
* A history of any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in mean Total Rhinoconjunctivitis Symptom Score (TRSS) | Between Baseline and approximately 25 weeks after randomisation

SECONDARY OUTCOMES:
Change from baseline in mean Total Rhinoconjunctivitis Symptom Score (TRSS) - all timepoints | Between Baseline and approximately 25 weeks after randomisation
Change from Baseline in mean Total Nasal Symptom Score (TNSS) | Aproximately 25 weeks after randomisation
Change from Baseline in mean Total Non Nasal Symptom Scores (TNNSS) | Approximately 25 weeks after randomisation
Number of Participants with Adverse Events as a Measure of Safety and tolerability | Approximately 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Piyush Patel, MD, Principal Investigator — Inflamax Research
Locations (5):
- Canada (5):
  - Kanata Allergy Services, Kanata, Ontario
  - KGK Synergize Inc, London, Ontario
  - Inflamax Research, Mississauga, Ontario
  - Taunton Health Centre, Oshawa, Ontario
  - Windsor Allergy Asthma Associates, Windsor, Ontario